CLINICAL TRIAL: NCT02160015
Title: A Phase 1 Study of Lenalidomide and Ibrutinib in Combination With Rituximab in Relapsed and Refractory CLL and SLL
Brief Title: Lenalidomide, Ibrutinib, and Rituximab in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma That Is Metastatic or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01157; NCI-2014-01157 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-00531; 2013-1342; 9540 (Other: MedStar Georgetown University Hospital); 9540 (Other: CTEP); P30CA051008 (NIH)
Record Dates: First submitted 2014-05-30; First posted 2014-06-10 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; ibrutinib; Lenalidomide; Magnetic Resonance Spectroscopy; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (lenalidomide, ibrutinib, rituximab) (Experimental): Patients receive rituximab IV on day 1 (up to 6 cycles), lenalidomide PO QD on days 1-21 (up to 12 cycles), and ibrutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECG on screening and CT scan or MRI, bone marrow biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Electrocardiogram; Drug: Ibrutinib; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Biological: Rituximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Electrocardiogram — Undergo ECG
  Other Names: ECG; EKG; Electrocardiograms
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with ibrutinib and rituximab in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma that has come back (relapsed), has not responded well to prior treatments (refractory), has spread to other parts of the body (metastatic), or cannot be removed by surgery. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving lenalidomide together with ibrutinib and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II doses of lenalidomide and ibrutinib for combination with rituximab in previously treated chronic lymphocytic leukemia and small lymphocytic lymphoma.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of lenalidomide, ibrutinib and rituximab in previously treated chronic lymphocytic leukemia and small lymphocytic lymphoma.

II. To describe any preliminary evidence of antitumor activity of the combination of lenalidomide, rituximab and ibrutinib in previously treated chronic lymphocytic leukemia and small lymphocytic lymphoma as defined by response rate, duration of response, and progression-free survival.

III. To observe and record anti-tumor activity.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive rituximab intravenously (IV) on day 1 (up to 6 cycles), lenalidomide orally (PO) once daily (QD) on days 1-21 (up to 12 cycles), and ibrutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo electrocardiogram (ECG) on screening and computed tomography (CT) scan or magnetic resonance imaging (MRI), bone marrow biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; previously treated, pathologically confirmed chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that requires as per the National Cancer Institute (NCI) Working Group Guidelines for the treatment of CLL; the diagnosis of CLL is defined by the presence of 5 x 10^9 clonal B-lymphocytes/L in the peripheral blood; clonality of the lymphocyte population is established with flow cytometry and the demonstration of the following surface markers: CD5, CD23, CD19, CD20 and the presence of either kappa or lambda immunoglobulins; the diagnosis of SLL may be made with the demonstration of < 5 x 10^9 clonal B-lymphocytes/L in the peripheral blood, with the clinical or radiographic features of enlarged lymph nodes or organomegaly, and the demonstration of SLL cells in the lymph node biopsy; institutional flow cytometry or immunohistochemistry must confirm CD20 antigen expression; patients may not have had a history of Richter's transformation
* No prior systemic therapy for CLL or SLL including chemotherapy or immunotherapy (e.g., monoclonal antibody-based therapy), radiation therapy, within 4 weeks of enrollment; no prior carmustine (BCNU) or mitomycin C within 6 weeks of enrollment; no radioimmunotherapy within a year of enrollment; no corticosteroids administered within 2 weeks prior to study entry, except for maintenance therapy (=< prednisone 20 mg daily or equivalent) for a non-malignant disease
* Patients may have had a prior autologous stem cell transplant; no prior history of allogeneic stem cell transplant
* Patients may have received prior lenalidomide as long as it has been at least two years since exposure and the patient may not have experienced a progression while receiving lenalidomide previously
* No Bruton's tyrosine kinase inhibitor at any point prior to enrollment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib, lenalidomide or rituximab or hypersensitivity to murine proteins or to any component of rituximab
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions if present should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow (involvement by SLL or CLL should be noted)
* No concomitant approved anti-cancer therapies or any investigational agents
* Patients with active or uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP) are excluded; patients who have transfusion-dependent thrombocytopenia or bleeding/coagulation disorders that may increase the risk of life-threatening bleeding are excluded
* Eastern Cooperative Oncology Group (ECOG) performance status must be < 2
* Patients with human immunodeficiency virus (HIV) infection are eligible, provided they meet the following:

  * No evidence of co-infection with hepatitis B or C
  * CD4+ cell count >= 400/mm^3
  * No evidence of resistant strains of HIV
* Patients with a prior diagnosis of CLL/SLL in central nervous system (CNS) are eligible only if the CNS disease has been treated; patients must be neurologically stable, without progressive symptoms while off of steroids and anti-convulsants; at least 28 days must have elapsed since CNS treatment, and the patient must have recovered from all associated toxicities of treatment; patients who have transfusion-dependent thrombocytopenia or bleeding/coagulation disorders that may increase the risk of life-threatening bleeding are excluded
* No evidence of active hepatitis B or C infections (hepatitis B surface antigen positive [HBsAg +], hepatitis B deoxyribonucleic acid [DNA] positive by polymerase chain reaction [PCR], or anti-hepatitis C virus [HCV] antibodies); hepatitis core antibody (HBcAb) seropositive patients that are HBsAg negative are eligible if they are closely monitored for evidence of active hepatitis B virus (HBV) infection by HBV DNA testing and receive suppressive therapy with lamivudine or other HBV suppressive therapy until 6 months after the last rituximab dose
* Patients must be non-pregnant and non-nursing; the effects of ibrutinib on the developing human fetus are unknown; for this reason and because B- cell receptor kinase inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for at least 3 days after discontinuation of ibrutinib, 28 days after discontinuation of lenalidomide, and 12 months after discontinuation of rituximab
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Contraception is recommended for 28 days prior to starting therapy, while participating in this study, during dose interruptions, and for at least 3 days after discontinuation of ibrutinib, 28 days after discontinuation of lenalidomide, and 12 months after discontinuation of rituximab
* No history of known human anti-chimeric antibody (HACA) positivity; this does not have to be checked prior to enrollment unless clinically indicated
* Life expectancy must be greater than 60 days
* No history of erythema multiforme, toxic epidermal necrolysis or Stevens-Johnson syndrome
* No history of uncontrolled seizures
* No autoimmune disorder that requires active immunosuppression
* No stroke or intracranial hemorrhage within the last 6 months
* No major surgery within 28 days prior to treatment; no minor surgery within 5 days prior to treatment
* No history of a congestive heart failure, myocardial infarction, unstable angina, uncontrolled arrhythmia, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification in the last 6 months
* No uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No prior malignancy with the exceptions listed below:

  * Malignancy treated with curative intent and with no evidence of active disease for more than 3 years prior to screening and felt to be at low risk (< 30%) for recurrence by the treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
* No use of warfarin or similar vitamin K antagonists
* No oral or intravenous corticosteroid use within 2 weeks prior to study entry
* Inhaled steroids are permitted
* Patients unable to swallow capsules, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption, such as malabsorption syndrome, resection of the small bowel, or poorly controlled inflammatory bowel disease affecting the small intestine are ineligible
* Patients should not receive growth factors or transfusions for at least 7 days prior to first dose of study drug, with the exception of pegylated G-CSF (pegfilgrastim) and darbopoeitin which require at least 14 days prior to screening and randomization
* Absolute neutrophil count > 750 cells/mcL (0.75 x 10^9/L)
* Platelet count > 50,000 cells/mcL (50 x 10^9/L)
* Hemoglobin > 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless Gilbert's syndrome or disease infiltration of the liver is present)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Creatinine clearance estimated (est.) glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 (Cockcroft-Gault)
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN
* A minimum organ function requirement may be waived if the malignancy being treated has involvement of the relevant organ

Exclusion Criteria:

* Chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 6 weeks prior to first administration of study treatment
* Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib
* Patients who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or patients who require continuous treatment with a strong CYP3A inhibitor
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or an infection requiring systemic antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; recent infections requiring systemic treatment need to have completed therapy > 14 days before the first dose of study drug
* Pregnant and breastfeeding women are excluded from this study; pregnant women are excluded in this study because ibrutinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ibrutinib, breastfeeding should be discontinued if the mother is treated with ibrutinib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are eligible; unless the patient's CD4 count is below the institutional lower limit of normal
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP) resulting in (or as evidenced by) declining platelet or hemoglobin (Hgb) levels within the 4 weeks prior to first dose of study drug
* Presence of transfusion-dependent thrombocytopenia
* Patients requiring daily corticosteroids at a prednisone equivalent of >= 20 mg daily should not be enrolled; if corticosteroids can be discontinued (or reduced to < 20 mg per day of prednisone or equivalent), the discontinuation or dose reduction should be done at least 7 days prior to first dose
* History of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
* Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Serologic status reflecting active hepatitis B or C infection; patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment; (PCR positive patients will be excluded)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the patient's safety, or put the study at undue risk
* Concomitant use of warfarin or other vitamin K antagonists
* Concurrent systemic immunosuppressant therapy other than corticosteroids (e.g., cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Major surgery within 4 weeks of first dose of study drug
* Unwilling or unable to participate in all required study evaluations and procedures
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the NCI/Child Pugh classification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2026-08-13 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of lenalidomide and ibrutinib with rituximab based on the maximum tolerated dose and the assessment of any clinically relevant toxicity | Up to 28 days
  Graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days following the last dose of ibrutinib
  Graded according to NCI CTCAE version 4.0. Descriptive statistics will be used in the analysis of all laboratory and safety parameters (adverse events, serious adverse events, adverse events leading to discontinuation, deaths) for all treated patients.
Overall response rate | From the start of the treatment until disease progression/recurrence or death, assessed up to 10 years
  The proportion of patients who achieve stable disease (SD) or a partial response (PR) or complete response (CR) will be reported with a 95% exact binomial confidence interval.
Complete response rates | Up to 10 years
  The proportion of patients who achieve CR will be reported with a 95% exact binomial confidence interval.
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed up to 10 years
Progression-free survival | Time from start of treatment to time of progression or relapse or death, whichever occurs first, assessed up to 10 years
  The progression-free survival will be evaluated using the methods of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Kieron Dunleavy, Principal Investigator — MedStar Georgetown University Hospital
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Hackensack University Medical Center, Hackensack, New Jersey